CLINICAL TRIAL: NCT06367439
Title: Examining the Effects of Virtual Reality Exercise on Mental Health Outcomes: A Randomized Controlled Trial
Brief Title: Examining the Effects of Virtual Reality Exercise on Mental Health
Acronym: UVIC VR Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Meta Platforms, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FN-10984
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Mental Health; Mood; Well-Being, Psychological; Physical Activity
Keywords: Virtual reality; Exergaming; Physical activity; Exercise
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will utilize a 10-week, two-arm, single-blinded, waitlist control, randomized controlled trial (RCT). Healthy adults (19-64 years) from the Victoria community participating in less than 75 minutes of vigorous physical activity per week will be randomized to either the Supernatural (SN) condition or the wait-list control (WLC) condition for a 10-week period.
Who Masked: Investigator
Masking Description: Single - Primary Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Exercise Condition (Experimental): Participants will complete a virtual reality (VR) exercise tutorial (Supernatural gameplay) and a Supernatural affect measurement workout (Flow or Boxing) in the Behavioural Medicine Lab (UVic). The tutorial will include watching Supernatural YouTube instructional videos, then completing a Supernatural training (~5-6 min), a 'getting started' low intensity Supernatural workout (~3 min), a low intensity Supernatural workout (~3 min), and a medium intensity Supernatural workout (~3 min). Participants will then complete the affect measurement medium intensity Supernatural workout (18-20 min). Participants will be provided a Virtual Reality headset (i.e., Meta Quest 3 headset) equipped with a Supernatural account for 10 weeks and will be instructed to participate in 75 minutes of medium intensity Supernatural physical activity per week which is equivalent to 75 minutes of vigorous physical activity (in line with the Canadian physical activity guidelines).
  Interventions: Behavioral: Virtual reality exercise condition
- Waitlist Control Condition (No Intervention): Participants will complete a control treadmill walk/run exercise session in the Behavioural Medicine Lab (30 min) that emulates the lab-based Supernatural exercise session (intervention condition). The treadmill run/walk will be the comparison condition for examining the effects of Supernatural exercise on mood and affect. First, participants will complete a 10 min treadmill orientation where they will walk for 3 min at 3 mph, walk for 3 min at 3.5 mph, walk/jog for 3 min at 4 mph, and walk for 1 min at 3 mph. Participants will then complete a 19.5-20 min treadmill walk/jog where they will complete a 1 min warmup at 3 mph, walk/jog for 17.5 min at 4 mph. Participants will then be asked to continue as they are for 10 weeks and will have the opportunity to bring home the Meta Quest 3 headset equipped with Supernatural for 10 weeks post-study.

INTERVENTIONS:
Behavioral: Virtual reality exercise condition — Participants will complete a virtual reality exercise (i.e., Supernatural) tutorial (YouTube instruction and in-headset gameplay instruction/practice) and will complete a 18-20 minute affect measurement medium intensity virtual reality exercise (i.e., Supernatural) session in the Behavioural Medicine Lab (UVic).
  Other Names: Baseline virtual reality exercise and measurement workout
  Arms: Virtual Reality Exercise Condition
Behavioral: Virtual reality exercise condition — Participants will be provided a virtual reality headset (Meta Quest 3 Headset) and subscription to a virtual reality exercise game (i.e., Supernatural) for 10 weeks. Participants will be instructed to participate in 75 minutes of medium intensity Supernatural physical activity (equivalent to 75 minutes of vigorous physical activity) per week in their own home.
  Other Names: 10 week virtual reality exercise program
  Arms: Virtual Reality Exercise Condition

SUMMARY:
The primary purpose of this investigation is to examine the efficacy of virtual reality (VR) exercise (Supernatural exergaming via Meta Platforms Technologies, LLC) for improving well-being (i.e., vitality) over a 10-week period. The secondary purpose is to examine the efficacy of VR exercise for improving depression mood symptoms, anxiety mood symptoms, and perceived cognitive functioning over a 10-week period, as well as short-term mood (post-exercise) and affective experiences during exercise. The tertiarty purpose of this study is to examine the efficacy of VR exercise for improving both physical activity behaviour and physical activity motivation (attitudes, capability, opportunity, intentions, behavioural regulation, habit, identity) over a 10-week period. Another tertiary purpose is to examine whether key motivational variables (e.g., attitudes, capability, opportunity, intentions, behavioural regulation, habit, identity) regarding Supernatural use explain variability in Supernatural use over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-64
* Living in the Greater Victoria area
* Have a stable Wi-Fi connection at home
* Experience no health constraints that limit moderate-to-vigorous physical activity participation as identified by the Physical Activity Readiness Questionnaire (PARQ+).
* Currently participating in less than 75 minutes of vigorous physical activity per week (as per Canadian physical activity guidelines)
* Be willing to travel into the Behavioural Medicine Lab on the UVic campus
* Be the only member of their household to participate in the study, past or present

Exclusion Criteria:

* If participant is flagged by the PARQ+ and is not cleared to participate in physical activity by their physician they are ineligible to participate
* Does not meet any of the above inclusion criteria

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Well-being: subjective vitality | Baseline, week 5, week 10
  Subjective vitality will be assessed using a six-item subjective vitality scale. Participants will respond to the six subjective vitality items on a seven point Likert-type scale anchored by 1 (not at all true) to 7 (very true). The six items will be mean scored (potential range 1-7), with higher scores reflecting higher subjective vitality and a more positive outcome.

SECONDARY OUTCOMES:
Depression and anxiety mood symptoms | Baseline, week 5, week 10
  Participants will respond to the 14-item Hospital Anxiety and Depression Scale, which includes a depression subscale (7 items) and an anxiety subscale (7 items). Participants will respond to the 14-items using a four point (0-3) Likert-type scale. The two subscales will be mean scored (potential range 0-3), with higher scores reflecting higher depression and anxiety and more negative outcomes.
Perceived cognitive function | Baseline, week 5, week 10
  Participants will respond to the organization (5 items) and strategic planning (7 items) subscales of the executive function index using a five point Likert-type scale anchored by 1 (Not at all) to 5 (Very much). The two subscales will be mean scored (potential range 1-5), with higher scores reflecting higher organization and strategic planning and more positive outcomes.
Short-term Mood | Pre (baseline) and post in-lab physical activity; through lab completion (2 hours).
  Participants will respond to the positive mood valence (2 items), calmness (2 items), and energy (2 items) sub-scales of the multidimensional mood questionnaire using a seven point Likert-type scale. The three subscales will be mean scored (potential range 0-6), with higher scores indicating a more positive mood (valence, calmness, energy) and a more positive outcome.
Core Affect Measure - Feeling Scale | Baseline (pre exercise session), at ~3.5 minute intervals during exercise (post song), and at 1.5 and 3 minutes post exercise). 8 measurements total
  Participants will complete a single item affect measure on an 11-point Likert-type scale anchored by -5 (very bad) to +5 (very good) to examine the affective response to exercise (Supernatural VR exercise or treadmill running). Higher scores will reflect more positive affective responses and a more positive outcome. Participants will be verbally prompted to respond to the scale during exercise (Supernatural VR exercise or treadmill exercise).
Core Affect Measure - Felt Arousal Scale | Baseline (pre exercise session), ~ at 3.5 minute intervals during exercise (post song), and at 1.5 and 3 minutes post exercise). 8 measurements total
  Participants will complete a single item arousal measure on a 6-point Likert-type scale anchored by 1 (low arousal) to 6 (high arousal). Participants will be verbally prompted to respond to the scale during exercise (Supernatural VR exercise or treadmill exercise).

OTHER OUTCOMES:
Perceived exertion | ~3.5 minute intervals (post song) during exercise. 5 measurements total.
  Using the modified Borg Rating of Perceived Exertion scale, participants will rate how hard they feel they are physically exerting themselves on a scale anchored by 0 (nothing at all) to 10 (very strong) during the exercise session (Supernatural VR exercise and treadmill running). Participants will be verbally prompted to respond to the scale during exercise.
Supernatural Target Accuracy | Once during in-lab Supernatural orientation (tutorial workout), and after each of the five songs completed during the in-lab Supernatural workout.
  Participants will receive a target accuracy score (i.e., number of targets successfully striked/punched) for each workout they complete. Scores range from 0 to 100%, with higher scores reflecting a more positive outcome.
Attitude towards physical activity | Baseline, week 5, week 10
  Participants will respond to three items assessing affective attitudes towards physical activity (boring-fun, unpleasant-pleasant, unenjoyable-enjoyable) and three items assessing instrumental attitudes towards physical activity (useless-useful, harmful-beneficial, unwise-wise), for the next five weeks. They will respond to the six items on a seven point Likert-type scale. The two subscales will be mean scored (potential range 1-7), with higher scores reflecting more positive affective attitudes and more positive instrumental attitudes towards physical activity and more positive outcomes.
Attitude towards Supernatural physical activity | Week 1, Week 5, Week 10
  Participants will respond to three items assessing affective attitudes towards Supernatural physical activity (boring-fun, unpleasant-pleasant, unenjoyable-enjoyable) and three items assessing instrumental attitudes towards Supernatural physical activity (useless-useful, harmful-beneficial, unwise-wise), for the next four/five weeks. They will respond to the six items on a seven point Likert-type scale. The two subscales will be mean scored (potential range 1-7), with higher scores reflecting more positive affective attitudes and more positive instrumental attitudes towards Supernatural physical activity and more positive outcomes.
Perceived opportunity for physical activity | Baseline, week 5, week 10
  Perceived opportunity to be regularly physically active over the next five weeks will be assessed using a three item scale. Participants will respond to the items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The three items will be mean scored (potential range 1-7), with higher scores indicating higher perceived opportunity for physical activity and a more positive outcome.
Perceived opportunity for Supernatural physical activity | Week 1, week 5, week 10
  Perceived opportunity to participate in regular Supernatural physical activity over the next four/five weeks will be assessed using an adapted three item scale. Participants will respond to the items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The three items will be mean scored (potential range 1-7), with higher scores indicating higher perceived opportunity for Supernatural physical activity and a more positive outcome.
Perceived capability for physical activity | Baseline, week 5, week 10
  Perceived capability for regular physical activity over the next five weeks will be assessed using a four item scale. Participants will respond to the four items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The four items will be mean scored (potential range 1-7), with higher scores indicating higher perceived capability for physical activity and a more positive outcome.
Perceived capability for Supernatural physical activity | Week 1, week 5, week 10
  Perceived capability for regular Supernatural physical activity over the next four/five weeks will be assessed using a four item scale. Participants will respond to the four items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The four items will be mean scored (potential range 1-7), with higher scores indicating higher perceived capability for Supernatural physical activity and a more positive outcome.
Intentions for physical activity behaviour | Baseline, week 5, week 10
  Participants will complete two items. First participants will report the number of minutes of moderate-to-vigorous physical activity they intend to complete in the next five weeks with a minimum score of 0 minutes and higher values reflecting a more positive outcome. Second, participants will report the strength of their desire to participate in regular physical activity over the next five weeks using a seven-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores (potential range 1-7) will reflect greater intention to participate in regular physical activity and a more positive outcome.
Intention for regular Supernatural physical activity behaviour | Week 1, week 5, week 10
  Participants will complete two items. First participants will report the number of minutes of medium intensity Supernatural physical activity they intend to complete in the next four/five weeks with a minimum score of 0 minutes and higher values reflecting a more positive outcome. Second, participants will report the strength of their desire to participate in regular Supernatural physical activity over the next four/five weeks using a seven-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores (potential range 1-7) will reflect greater intention to participate in regular physical activity and a more positive outcome.
Behavioural regulation of physical activity behaviour | Baseline, week 5, week 10
  Participants will respond to the 14-item physical activity regulation scale using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The 14-item measure includes four subscales, which are proactive regulation (4 items), reactive regulation (4 items), social monitoring (3 items), and self-monitoring (3 items).The four subscales will be mean scored (potential range 1-7), with higher scores indicating higher levels of physical activity behaviour regulation and a more positive outcome.
Behavioural regulation of Supernatural physical activity | Week 1, week 5, week 10
  Participants will respond to the 14-item physical activity regulation scale adapted for Supernatural physical activity using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The 14-item measure includes four subscales, which are proactive regulation (4 items), reactive regulation (4 items), social monitoring (3 items), and self-monitoring (3 items).The four subscales will be mean scored (potential range 1-7), with higher scores indicating higher levels of Supernatural physical activity behaviour regulation and a more positive outcome.
Physical activity habit | Baseline, week 5, week 10
  Participants will complete the four item self-report behavioural automaticity index. Participants will respond to four items on a five point Likert-type scale anchored by 1 (strongly disagree) to 5 (strongly agree). The four items will be mean scored (potential range 1-5), with higher scores reflecting a stronger physical activity habit and a more positive outcome.
Supernatural physical activity habit | Week 1, week 5, week 10
  Participants will complete the four item self-report behavioural automaticity index, adapted for Supernatural physical activity. Participants will respond to four items on a five point Likert-type scale anchored by 1 (strongly disagree) to 5 (strongly agree). The four items will be mean scored (potential range 1-5), with higher scores reflecting a stronger Supernatural physical activity habit and a more positive outcome.
Physical activity identity | Baseline, week 5, week 10
  Physical activity identity will be assessed using the three item self-identity subscale of the exercise identity scale. Participants will respond to the three items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The three items will be mean scored (potential range 1-7), with higher score reflecting a greater physical activity self-identity and a more positive outcome.
Supernatural physical activity identity | Week 1, week 5, week 10
  Supernatural physical activity identity will be assessed using an adapted three item self-identity subscale of the exercise identity scale. Participants will respond to the three items using a seven point Likert-type scale anchored by 1 (strongly disagree) to 7 (strongly agree). The three items will be mean scored (potential range 1-7), with higher score reflecting a greater Supernatural physical activity self-identity and a more positive outcome.
Physical activity behaviour | Baseline, week 5, week 10
  In reference to the past five weeks, participants will report the number of times per week (on average) they engaged in mild, moderate, and vigorous physical activity using the Godin Leisure Time Exercise Questionnaire, and the average duration of mild, moderate, and vigorous physical activity sessions. The researchers will create an indicator of average weekly moderate-to-vigorous physical activity minutes (in past 5 weeks) for each participant using the following equation: (number of moderate bouts x average minutes per bout) + (number of vigorous bouts x average minutes per bout). The scores will have a minimum value of 0 minutes, with more minutes indicating greater participation in moderate-to-vigorous physical activity and a more positive outcome.
Supernatural physical activity behaviour | Week 1, Week 5, week 10
  In reference to the past one/four/five weeks, participants will report the number of times per week (on average) they engaged in low, medium, and high intensity Supernatural physical activity using the Godin Leisure Time Exercise Questionnaire, and the average duration of the low, medium, and high intensity Supernatural physical activity sessions. The researchers will create an indicator of average weekly medium-high intensity Supernatural physical activity minutes for each participant using the following equation: (number of medium bouts x average minutes per bout) + (number of high bouts x average minutes per bout). The scores will have a minimum value of 0 minutes, with more minutes indicating greater participation in Supernatural physical activity and a more positive outcome.
Weekly Supernatural Physical Activity Behaviour | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10
  Participants in the Supernatural condition will log their Supernatural VR physical activity (intensity and duration for each day of the week) at the end of each week. Scores will have a minimum value of 0 minutes, with more minutes indicating greater participation in Supernatural physical activity and a more positive outcome.
Direct assessment of Supernatural physical activity behaviour | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10
  The Meta Quest Move application (within Meta Quest 3 headset) estimates the amount of calories expended and 'move minutes' for each application in the headset. The calories expended and move minutes (within a particular time frame) in Supernatural will be extracted from the Meta Quest Move application for each participant. Meta Quest Move does underestimate the number of calories expended during a bout of physical activity and will therefore represent a proxy measure for Supernatural engagement time. A total score for calories burned and 'move minutes' will be recorded for each week of the study, with minimum values of 0 minutes and 0 calories and more minutes and calories expended indicating greater participation in Supernatural physical activity and a more positive outcome.
Direct assessment of physical activity behaviour | Baseline and Week 10
  Accelerometers (wGT3X-BT ActiGraph) will provide direct assessments of participants' moderate-to-vigorous physical activity. Participants will wear the accelerometer for seven days at baseline and seven days post-week 10. The scores will have a minimum value of 0 minutes with more minutes will indicate greater participation in moderate-to-vigorous physical activity and a more positive outcome.
Feasibility and Acceptability of Supernatural and the Meta Quest 3 headset | Week 10
  Participants in the Supernatural condition will complete 9 items regarding the feasibility and acceptability of the Supernatural VR exercise game and the Meta Quest 3 headset. Participants will respond to each item on a five point Likert scale anchored by 1 (strongly disagree) to 5 (strongly agree). The 9 items will be mean scored (potential range 1-5), with higher scores indicating higher levels of feasibility and acceptability for both Supernatural VR exercise game and the Meta Quest 3 and a more positive outcomes. Items were derived from a previous Feasibility study. A sub-group of participants in the Supernatural condition will participate in exit interviews regarding the feasibility and acceptability of Supernatural VR exercise game and the Meta Quest 3 headset.
Supernatural usability | Week 10
  Participants in the Supernatural condition will complete an adapted 10-item system usability scale for the Supernatural VR exercise game, responding to each item on a five point Likert scale anchored by 1 (strongly disagree) to 5 (strongly agree).The 10-items will be mean scored (potential range 1-5), with higher scores indicating higher levels of Supernatural usability and a more positive outcome. A sup-group of participants in the Supernatural condition will participate in exit interviews regarding the usability of the Supernatural VR exercise game.
Meta Quest 3 headset usability | Week 10
  Participants in the Supernatural condition will complete an adapted 10-item system usability scale for the Meta Quest 3 headset, responding to each item on a five point Likert scale anchored by 1 (strongly disagree) to 5 (strongly agree).The 10-items will be mean scored (potential range 1-5), with higher scores indicating higher levels of Meta Quest 3 usability and a more positive outcome. A sub-group of participants in the Supernatural condition will participate in exit interviews regarding the usability of the Meta Quest 3 headset.
Personality | Week 5
  Participants will respond to the neuroticism (12 items), extraversion (12 items), and conscientiousness (12 items) subscales in the five factor inventory. Participants will respond to the 36 personality related items on a five point Likert-type scale anchored by 0 (strongly disagree) to 4 (strongly agree). Each subscale will be mean scored (potential range 0-4), with higher scores reflecting a higher degree of the personality trait.
Physical Activity Environment | Week 10
  The environmental module of the International Physical Activity Prevalence Study (IPS) will be used to assess a participants environment for walking and bicycling ability . Participants will be able to respond 17 items on a four point Likert-type scale anchored by 1 (strongly disagree) to 4 (strongly agree). Items will be mean scored (potential range 1 to 4) with higher scores reflecting a more favourable environment for physical activity participation.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — Lab Director and Professor
Locations (1):
- Behavioural Medicine Lab, Victoria, British Columbia, Canada

REFERENCES:
- [Background] Borg, G. (1998). Borg's perceived exertion and pain scales. Human Kinetics.
- [Background] Courneya, K. S. (1994). Predicting repeated behavior from intention: The issue of scale correspondence. Journal of Applied Social Psychology, 24(7), 580-594. https://doi.org/10.1111/j.1559-1816.1994.tb00601.x
- [Background] Courneya KS, Jones LW, Rhodes RE, Blanchard CM. Effects of different combinations of intensity categories on self-reported exercise. Res Q Exerc Sport. 2004 Dec;75(4):429-33. doi: 10.1080/02701367.2004.10609176. No abstract available. PMID 15673042
- [Background] Costa, P. T., & McCrae, R. R. (1992). Revised neo personality inventory and Neo Five-Factor Inventory. Research Psychologists Press.
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Hardy, C. J., & Rejeski, W. J. (1989). Not what, but how one feels: The measurement of affect during exercise. Journal of Sport & Exercise Psychology, 11, 304-317.
- [Background] IPAQ. (2004). International physical activity prevalence study environmental survey module. Retrieved August 10 from http://www-rohan.sdsu.edu/faculty/sallis/IPAQIPS.pdf
- [Background] Lithopoulos A, Zhang CQ, Williams DM, Rhodes RE. Development and Validation of a Two-component Perceived Control Measure. Ann Behav Med. 2023 Feb 4;57(2):175-184. doi: 10.1093/abm/kaac033. PMID 35849341
- [Background] Rhodes RE, Courneya KS. Investigating multiple components of attitude, subjective norm, and perceived control: an examination of the theory of planned behaviour in the exercise domain. Br J Soc Psychol. 2003 Mar;42(Pt 1):129-46. doi: 10.1348/014466603763276162. PMID 12713760
- [Background] Rhodes, R. E., & Courneya, K. S. (2004). Differentiating motivation and control in the Theory of Planned Behavior. Psychology, Health, and Medicine, 9(2), 205-215. https://doi.org/10.1080/13548500410001670726
- [Background] Rhodes RE, Lithopoulos A. The Physical Activity Regulation Scale: Development and validity testing. Health Psychol. 2023 Jun;42(6):378-387. doi: 10.1037/hea0001283. PMID 37227880
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Spinella M. Self-rated executive function: development of the executive function index. Int J Neurosci. 2005 May;115(5):649-67. doi: 10.1080/00207450590524304. PMID 15823930
- [Background] Svebak, S., & Murgatroyd, S. (1985). Metamotivational dominance: A multimethod validation of reversal theory constructs. Journal of Personality and Social Psychology, 48(1), 107-116.
- [Background] Wilhelm, P., & Schoebi, D. (2007). Assessing mood in daily life: Structural validity, sensitivity to change, and reliability of a short-scale to measure three basic dimensions of mood. European Journal of Psychological Assessment, 23(4), 258-267. https://doi.org/10.1027/1015-5759.23.4.258
- [Background] Wilson, P. M., & Muon, S. (2008). Psychometric properties of the Exercise Identity Scale in a university sample. International Journal of Sport and Exercise Psychology, 6(2), 115-131. https://doi.org/10.1080/1612197X.2008.9671857
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Anderson DF, Cychosz CM. Development of an exercise identity scale. Percept Mot Skills. 1994 Jun;78(3 Pt 1):747-51. doi: 10.1177/003151259407800313. PMID 8084685
- [Background] Bostic, T. J., Rubio, D. M., & Hood, M. (2000). A validation of the subjective vitality scale using structural equation modelling. Social Indicators Research, 52(3), 313-324. https://doi.org/10.1111/j.1541-0072.1977.tb01338.x
- [Background] Cox A, Rhodes RE. Increasing Physical Activity in Empty Nest and Retired Populations Online: A Randomized Feasibility Study. J Aging Phys Act. 2023 Jun 1;31(6):909-922. doi: 10.1123/japa.2022-0285. Print 2023 Dec 1. PMID 37263598
- [Background] Peres, S. C., Pham, T., & Phillips, R. (2013). Validation of the system usability scale (sus): SUS in the wild. Proceedings of the Human Factors and Ergonomics Society, 1, 192-196. https://doi.org/10.1177/1541931213571043